CLINICAL TRIAL: NCT04151459
Title: Effect of Laparoscopic Sleeve Gastrectomy (LSG) on Live Birth Rate of Offspring in Polycystic Ovarian Syndrome (PCOS) Patients With Severely Obese
Brief Title: Effect of Metabolic Surgery on Live Birth Rate of Offspring in Obesity Polycystic Ovarian Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2018]048
Record Dates: First submitted 2019-10-15; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Polycystic Ovary Syndrome; Severe Obesity; Laparoscopic Sleeve Gastrectomy
Keywords: Polycystic Ovary Syndrome; Severe Obesity; Laparoscopic Sleeve Gastrectomy; Live Birth Rate
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity, Morbid | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic sleeve gastrectomy (Experimental): Laparoscopic sleeve gastrectomy on severe obesity PCOS patients
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Use Metformin for 3 months to treat PCOS
  Other Names: Glucophage

SUMMARY:
This is a experimental study, which subjects are obese PCOS patients requiring LSG surgery. Aim to investigate the effects of LSG surgery in PCOS patients whether increases the live birth rate of the offspring.

DETAILED DESCRIPTION:
The investigators designed a single center small sample exploratory study to clear the therapeutic effects of laparoscopic sleeve gastrectomy on live birth rate improvements of overweight/obese PCOS patients. The investigators plan to enroll 18 patients. Inclusion criteria: 1) Patients who are aged from 18 to 45, not menopause;2) have PCOS which is diagnosed according to 2003 Rotterdam criteria; 3) have been treated with behavioral and drugs intervention for 3 months but are ineffective; 4) have steady or steady weight gain over 5 years, BMI>35kg/m2, or BMI>30kg/m2 with one of the metabolic disorders such as impaired glucose tolerance, cardiovascular disease, fatty liver, lipid metabolism disorders, sleep apnea syndrome.

Patients with serious complications (cardiovascular events and recent significant liver, kidney or lung disease within 3 months); high blood pressure (>160/100mmHg); active infection; secondary diabetes; pregnancy; alcohol abuse; surgical contraindications are excluded.

Then the investigators plan to perform laparoscopic sleeve gastrectomy . Before and after the intervention, the blood samples would be collected to detect blood glucose, insulin, lipid profile, sex hormones, blood chemistry for liver and kidney function, hsCRP etc., as well as the anthropometric measurement and image examinations. All patients are followed up every 3 months until the end of the program. All patients receive MRI plain scan of upper and lower abdomen, oral glucose tolerance test (OGTT) and insulin, C-peptide releasing test again every 6 months after the operation. One year after the operation, patients would be evaluated whether they are suitable for pregnancy preparation and record the pregnancy mode. After pregnancy, various indicators would be closely monitored, including maternal vitamin and trace element levels.The birth of children and the live birth rate would be recorded.

The investigators will compare the data and finally identify the treatment effect of laparoscopic sleeve gastrectomy on overweight/obese PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

- aged from 18 to 45, not menopause have PCOS which is diagnosed according to 2003 Rotterdam criteria have been treated with behavioral and drugs intervention for 3 months but are ineffective have steady or steady weight gain over 5 years, BMI>35kg/m2, or BMI>30kg/m2 with one of the metabolic disorders such as impaired glucose tolerance, cardiovascular disease, fatty liver, lipid metabolism disorders, sleep apnea syndrome

Exclusion Criteria:

- Except for serious complications (cardiovascular events and recent significant liver, kidney or lung disease within 3 months) high blood pressure (>160/100mmHg) active infection secondary diabetes pregnancy alcohol abuse surgical contraindications

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Improvement of metabolic surgery on live birth rate of offspring in obesity PCOS patients. | up to 3 years
  To record the offspring production and live birth rate of obesity PCOS patients after metabolic surgery

SECONDARY OUTCOMES:
Effect of metabolic surgery on ovulation rate and pregnancy rate of PCOS patients | up to 3 years
  To compare the ovulation rate and pregnancy of obesity PCOS patient with metabolic surgery or not
Effects of metabolic surgery on intestinal flora of PCOS patients and progeny. | up to 3 years
  To compare the intestinal flora of PCOS patients after metabolic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Study Chair — RenJi Hospital Department of Endocrinology and Metabolism
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li R, Zhang Q, Yang D, Li S, Lu S, Wu X, Wei Z, Song X, Wang X, Fu S, Lin J, Zhu Y, Jiang Y, Feng HL, Qiao J. Prevalence of polycystic ovary syndrome in women in China: a large community-based study. Hum Reprod. 2013 Sep;28(9):2562-9. doi: 10.1093/humrep/det262. Epub 2013 Jun 27. PMID 23814096
- [Background] Jarrett BY, Lujan ME. Impact of hypocaloric dietary intervention on ovulation in obese women with PCOS. Reproduction. 2017 Jan;153(1):R15-R27. doi: 10.1530/REP-16-0385. PMID 27799625
- [Background] Behboudi-Gandevani S, Ramezani Tehrani F, Rostami Dovom M, Farahmand M, Bahri Khomami M, Noroozzadeh M, Kabir A, Azizi F. Insulin resistance in obesity and polycystic ovary syndrome: systematic review and meta-analysis of observational studies. Gynecol Endocrinol. 2016;32(5):343-53. doi: 10.3109/09513590.2015.1117069. Epub 2016 Jan 6. PMID 27052492
- [Background] Skubleny D, Switzer NJ, Gill RS, Dykstra M, Shi X, Sagle MA, de Gara C, Birch DW, Karmali S. The Impact of Bariatric Surgery on Polycystic Ovary Syndrome: a Systematic Review and Meta-analysis. Obes Surg. 2016 Jan;26(1):169-76. doi: 10.1007/s11695-015-1902-5. PMID 26431698
- [Background] Niu Z, Lin N, Gu R, Sun Y, Feng Y. Associations between insulin resistance, free fatty acids, and oocyte quality in polycystic ovary syndrome during in vitro fertilization. J Clin Endocrinol Metab. 2014 Nov;99(11):E2269-76. doi: 10.1210/jc.2013-3942. Epub 2014 Apr 2. PMID 24694334
- [Background] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830